CLINICAL TRIAL: NCT01155453
Title: A Phase Ib, Open-label, Multi-center, Dose-escalation Study of Oral BKM120 in Combination With Oral GSK1120212 in Adult Patients With Selected Advanced Solid Tumors.
Brief Title: A Study to Investigate Safety, Pharmacokinetics (PK) and Pharmacodynamics (PD) of BKM120 Plus GSK1120212 in Selected Advanced Solid Tumor Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBKM120B2101; 2009-017157-35 (EudraCT Number)
Record Dates: First submitted 2010-06-17; First posted 2010-07-01 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2016-06

CONDITIONS: Advanced and Selected Solid Tumors
Keywords: BKM120; RAS RAF mutations,; triple negative breast cancer,; pancreatic cancer,; PI3K inhibitor,; MEK inhibitor
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Pancreatic Neoplasms | interventions — NVP-BKM120; trametinib

ARMS (4):
- BKM120 + GSK1120212 DE (Experimental): Dose Escalation
  Interventions: Drug: BKM120; Drug: GSK1120212
- BKM120 + GSK1120212 NSCLC patients (Experimental): Advanced RAS or BRAF mutant NSCLC patients
  Interventions: Drug: BKM120; Drug: GSK1120212
- BKM120 + GSK1120212 ovarian cancer patients (Experimental): Advanced RAS or BRAF mutant ovarian cancer patients
  Interventions: Drug: BKM120; Drug: GSK1120212
- BKM120 + GSK1120212 pancreatic cancer patients (Experimental): Advanced RAS or BRAF mutant pancreatic cancer patients
  Interventions: Drug: BKM120; Drug: GSK1120212

INTERVENTIONS:
Drug: BKM120
Drug: GSK1120212

SUMMARY:
This is an open label, dose finding, phase Ib clinical trial to determine the maximum tolerated dose (MTD) and /or recommended phase II dose (RP2D) and schedule for the PI3K (Phosphatidylinositol 3-Kinase) inhibitor BKM120 given in combination with the MEK inhibitor GSK1120212 in patients with selected, advanced solid tumors. The focus will be on tumors with RAS/RAF mutations and on triple negative breast cancer.

Both study drugs will be administered once daily orally on a continuous schedule, a treatment cycle is defined as 28 days.

Cohorts of at least 3 and up to a maximum of 6 patients eligible for the dose-determining set will be enrolled per dose combination below the MTD. The MTD is defined as the highest drug dosage not causing in the first cycle of treatment medically unacceptable, dose-limiting toxicity (DLT) in more than 33% of the treated patients.. At least 12 patients will be required at MTD and 6 patients at RP2D level to allow the evaluation of the combination's safety and pharmacokinetics or pharmacodynamics.

Upon declaration of MTD and/or RP2D, patients will be enrolled to an expansion part of the study, to further assess safety, as well as to learn more about the efficacy of the study drug combination.

* Expansion Arm 1 will consist of approximately 15 patients with RAS or BRAF mutant advanced NSCLC
* Expansion Arm 2 will consist of approximately 15 patients with RAS or BRAF-mutant ovarian cancer
* Expansion Arm 3 will consist of approximately 15 patients with RAS or BRAF-mutant pancreatic cancer

ELIGIBILITY:
Inclusion Criteria:

* histologically/ cytologically confirmed, advanced non resectable solid tumors
* Measurable or non-measurable, but evaluable disease as determined by RECIST 1.0

Exclusion Criteria:

* Patients with primary Central Nervous System (CNS) tumor or CNS tumor involvement.
* Clinically manifested diabetes mellitus - Unacceptable ocular/retinal conditions

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2010-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and/or recommended phase II dose (RP2D) and schedule of BKM120+GSK1120212 | in average 1 year

SECONDARY OUTCOMES:
Measure the number of Adverse Event and laboratory values that fall outside of pre-determined ranges as a measure of Safety and tolerability of the oral combination of BKM120 and GSK1120212 | in average 1 year
Determine the single and multiple dose pharmacokinetics of BKM120 and GSK1120212 in measurement of the plasma concentration profiles of BKM120 and GSK1120212 | Assessed during the first Cycle (28 days) of treatment
Preliminary anti-tumor activity of the combination | Assessed every 8 weeks of treatment
Treatment-induced PI3K and MEK/ERK(Mitogen-activated protein kinase /extracellular-signal-regulated kinases) pathway signaling inhibition and evidence of biological activity in tumor and skin | Assessed every 2 weeks during the first cycle, then every 4 weeks
Molecular status (genetic alterations, protein expression and/or activation) of markers related to PI3K and ERK signaling in tumor tissue and blood and investigate their potential relationship to clinical responses | Assessed at baseline (pre-treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- United States (2):
  - University of California at Los Angeles Div. of Hematology/Oncology, Los Angeles, California
  - University of Texas/MD Anderson Cancer Center Dept of MD Anderson (8), Houston, Texas
- Novartis Investigative Site, Leuven, Belgium
- Novartis Investigative Site, Toronto, Ontario, Canada
- Spain (2):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
- Novartis Investigative Site, Bellinzona, Switzerland

REFERENCES:
- See also: Results for CBKM120B2101 on the Novartis Clinical Trial website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13963